CLINICAL TRIAL: NCT02960243
Title: Left, Right, or Bilateral Thalamic Deep Brain Stimulation for Voice Tremor: A Prospective, Randomized, Double-Blinded Trial
Brief Title: Deep Brain Stimulation for Voice Tremor: Left, Right, or Both Hemispheres?
Acronym: EVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Honey, Neurosurgeon, Professor of Surgery (Neurosurgery), Director of Surgical Centre for Movement Disorders, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H16-01694
Record Dates: First submitted 2016-11-05; First posted 2016-11-09 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Essential Voice Tremor; Deep Brain Stimulation; Essential Tremor; Laryngeal Diseases; Action Tremor; Tremor, Nerve
Keywords: Deep Brain Stimulation; Laryngeal Motor Cortex; Essential Voice Tremor; Essential Tremor
MeSH Terms: conditions — Essential Tremor; Laryngeal Diseases; Tremor | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bilateral Thalamic Vim OFF (Sham Comparator): Participants with bilateral thalamic DBS will be tested four times over 90 minutes. The four tests will include the following in a randomized, double-blinded order:
  First test: both stimulators on for 15 minutes Second test: left stimulator off, right stimulator on for 15 minutes Third test: left stimulator on, right stimulator off for 15 minutes Fourth test: both stimulators off for 15 minutes
  In between switching to each test, there will be a 5 minute washout period.
  Interventions: Device: Deep Brain Stimulation
- Left Thalamic Vim ON (Experimental): Participants with bilateral thalamic DBS will be tested four times over 90 minutes. The four tests will include the following in a randomized, double-blinded order:
  First test: both stimulators on for 15 minutes Second test: left stimulator off, right stimulator on for 15 minutes Third test: left stimulator on, right stimulator off for 15 minutes Fourth test: both stimulators off for 15 minutes
  In between switching to each test, there will be a 5 minute washout period.
  Interventions: Device: Deep Brain Stimulation
- Right Thalamic Vim ON (Experimental): Participants with bilateral thalamic DBS will be tested four times over 90 minutes. The four tests will include the following in a randomized, double-blinded order:
  First test: both stimulators on for 15 minutes Second test: left stimulator off, right stimulator on for 15 minutes Third test: left stimulator on, right stimulator off for 15 minutes Fourth test: both stimulators off for 15 minutes
  In between switching to each test, there will be a 5 minute washout period.
  Interventions: Device: Deep Brain Stimulation
- Bilateral Thalamic Vim ON (Experimental): Participants with bilateral thalamic DBS will be tested four times over 90 minutes. The four tests will include the following in a randomized, double-blinded order:
  First test: both stimulators on for 15 minutes Second test: left stimulator off, right stimulator on for 15 minutes Third test: left stimulator on, right stimulator off for 15 minutes Fourth test: both stimulators off for 15 minutes
  In between switching to each test, there will be a 5 minute washout period.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — * DBS System Medtronic
  * DBS programming settings will be set to maximally alleviate limb tremor, primary reason for referral
  * These settings will be used to evaluate effects of voice tremor as well
  Other Names: DBS

SUMMARY:
Deep Brain Stimulation (DBS) is the gold standard treatment for Essential Tremor (ET). ET is a movement disorder which causes the arms, feet, fingers, head or voice to involuntarily shake. The DBS surgical procedure involves implanting an electrode deep within the brain which blocks damaging signals that cause the tremor. Essential Voice Tremor (EVT) is the vocal manifestation of ET and a number of individuals have both ET and EVT, and when these patients are implanted for their ET, their EVT symptoms are often also mitigated. This study aims to quantify the effects of DBS on EVT by testing on these ET+EVT patients. In addition to this, we hope to determine which hemisphere of the brain is responsible for larynx control: left or right.

DETAILED DESCRIPTION:
Essential Tremor (ET) is the most common movement disorder in adults, affecting approximately 5% of individuals over the age of 65. Of this 5%, roughly 20% of these patients suffer from Essential Voice Tremor (EVT): the phonatory manifestation of ET. Patients with EVT lose their ability to speak due to a tremor in the muscles of the larynx, pharynx, palate, and tongue. Because of this, an individual's quality of life is limited because they can no longer communicate effectively.

The purpose of this study is to quantify to what degree Deep Brain Stimulation improves Essential Voice Tremor. In addition to this, we hope to examine which brain hemisphere is responsible for these positive results: right, left, or both, in a prospective, randomized, double-blinded manner. By finding out more about the subcortical control underpinning speech, we will be able to improve our treatments and understanding of EVT and other neurological speech disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participant has been implanted with the DBS for ET
* Participant has significant voice tremor as determined by our laryngology/speech-language pathology team

Exclusion Criteria:

* Participant does not have history of aphasia or other speech/language deficits
* Participant does not have history of stroke or multiple sclerosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
The Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) | At the end of each trial period, typically 15 minutes after change in stimulation settings
  Patients will be asked to read a voice protocol designed to elicit voice tremor symptoms. This will be conducted at the end of every trial arm with a patient sitting in a rest position without moving upper or lower limbs.

SECONDARY OUTCOMES:
Voice Tremor Severity | Measured every 3 minutes for 15 minutes
  At the end of the study, the kinetics of voice tremor and limb tremor will be analyzed to determine if there are any similarities or differences in the time course to deterioration

CONTACTS AND LOCATIONS:
Locations (1):
- The Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Simonyan K, Ostuni J, Ludlow CL, Horwitz B. Functional but not structural networks of the human laryngeal motor cortex show left hemispheric lateralization during syllable but not breathing production. J Neurosci. 2009 Nov 25;29(47):14912-23. doi: 10.1523/JNEUROSCI.4897-09.2009. PMID 19940187
- [Result] Mandat T, Koziara H, Rola R, Bonicki W, Nauman P. Thalamic deep brain stimulation in the treatment of essential tremor. Neurol Neurochir Pol. 2011 Jan-Feb;45(1):37-41. doi: 10.1016/s0028-3843(14)60058-x. PMID 21384292
- [Result] Koller WC, Lyons KE, Wilkinson SB, Troster AI, Pahwa R. Long-term safety and efficacy of unilateral deep brain stimulation of the thalamus in essential tremor. Mov Disord. 2001 May;16(3):464-8. doi: 10.1002/mds.1089. PMID 11391740